CLINICAL TRIAL: NCT01657188
Title: Effects of Adaptive Servoventilation in Patients With Systolic Heart Failure and Sleep-Disordered Breathing
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Olaf Oldenburg, Senior cardiologist, Ruhr University of Bochum
Other Study IDs: HDZNRW_KA_001_OO
Record Dates: First submitted 2012-07-27; First posted 2012-08-06 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Heart Failure, Congestive; Sleep Apnea Syndromes; Adaptive Servoventilation
Keywords: Heart failure, congestive; Sleep apnea syndromes; Adaptive servoventilation; Prognosis; Cheyne-Stokes respiration
MeSH Terms: conditions — Heart Failure; Sleep Apnea Syndromes; Cheyne-Stokes Respiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart failure, sleep-disordered breathing: Patients with stable heart failure NYHA ≥ II, EF ≤ 45% with or without central sleep apnea (apnea-hypopnea index ≥ 15/h) with or without adaptive servoventilation
  Interventions: Device: Cheyne-Stokes respiration by adaptive servoventilation

INTERVENTIONS:
Device: Cheyne-Stokes respiration by adaptive servoventilation

SUMMARY:
Prospective, follow-up registry of heart failure patients with or without sleep-disordered breathing (SDB). To test the hypothesis that treatment of nocturnal central sleep apnea with Cheyne-Stokes respiration by adaptive servoventilation (ASV) improves symptoms, cardiac performance and event-free survival.

DETAILED DESCRIPTION:
The study is intended to investigate therapeutic effects of adaptive servoventilation in patients with sleep-disordered breathing and chronic heart failure. These effects include short-/long-term effects on

* symptoms and quality of life
* physical and cardiac performance (6min walking test, cardiopulmonary exercise testing)
* echocardiographic parameters
* arrhythmias
* NT-proBNP
* Respiratory stability (blood gases, rebreathing test, VE/VCO2-slope in cardiopulmonary exercise testing)
* Compliance with ASV therapy
* Event free survival (death, heart transplantation, assist device implantation)

All of these data are also obtained in patients who basically meet the inclusion criteria but in whom sleep-disordered breathing was excluded by means of cardiorespiratory polygraphy or polysomnography and in patients with sleep-disordered breathing who do not undergo adaptive servoventilation for various reasons.

ELIGIBILITY:
Inclusion Criteria:

* Stable heart failure NYHA ≥ II
* EF ≤ 45%
* without sleep-disordered breathing (apnea-hypopnea-index <5/h) and those with moderate to severe central sleep apnea (apnea-hypopnea index ≥ 15/h) with or without adaptive servoventilation therapy

Exclusion Criteria:

* Cardiac resynchronization or pacemaker implantation within the last 6 months
* Significant COPD with an forced expiratory one-second capacity relative to vital capacity (FEV1/VC)< 70% (GOLD III)
* Respiratory insufficiency requiring long-term oxygen therapy
* Daytime hypercapnia at rest (pCO2 > 45 mmHg)
* Current ventilation therapy
* Cardiac surgery, PCI, myocardial infarction, unstable angina, TIA or stroke within 12 weeks prior to randomization
* Acute myocarditis within 6 months prior to randomization
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of a university hospital
Sampling Method: Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2009-05; Primary Completion 2016-02 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Influence of adaptive servoventilation on heart failure parameters including event free survival | Time frame for event free survival analysis is up to 8 years
  This prospective registry includes heart failure patients with or without accompanied sleep-disordered breathing and investigates its influence on symptoms, cardiac function and performance, quality of life and outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Oldenburg, M.D., Principal Investigator — Heart and Diabetes Center North Rhine-Westphalia, Ruhr University Bochum
Locations (1):
- Department of Cardiology, Heart and Diabetes Center North Rhine-Westphalia, Ruhr University Bochum, Bad Oeynhausen, Germany